CLINICAL TRIAL: NCT00632957
Title: Center for the Biologic Basis of Oral/Systemic Diseases Project 5: Oral Infections: Dietary Regulation of Local and Systemic Inflammatory Responses.
Brief Title: Oral Infections: Dietary Regulation of Local and Systemic Inflammatory Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Dr. Jeff L. Ebersole, PI, Center for Oral Health Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UK IRB # 04-0339-F1V; P20RR020145-04 (NIH)
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Periodontal Attachment Loss
MeSH Terms: conditions — Periodontal Attachment Loss | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Active Comparator)
  Interventions: Dietary Supplement: Omega-3 Fatty acid (with SRP or OHI)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty acid (with SRP or OHI) — 1000mg capsules three times daily, duration 28 weeks.
  Arms: Fish oil
Dietary Supplement: Placebo — corn/soybean oil capsules 1g/three times daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that dietary n-3 PUFA will have a beneficial effect on systemic and local markers of inflammation when combined with traditional, non-surgical periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age, male or female
2. At least 20 natural teeth present at the time of periodontal examination
3. Be diagnosed with severe, chronic periodontitis;
4. Be willing to participate in the study

Exclusion Criteria:

1. <18 years of age
2. Less than 20 natural teeth present at time of periodontal examination
3. Unable or unwilling to provide informed consent or follow study protocol
4. Systemic conditions including diabetes mellitus and any cardiovascular condition that would require premedication prior to dental treatment
5. Use of systemic antibiotics within the last 3 months
6. Pregnancy as diagnosed by administered pregnancy test.
7. You are nursing a baby.
8. Are allergic to fish or fish products.
9. You are taking any other medications, such as dietary supplements, that could affect the outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
clinical attachment loss | baseline, 8, 16, 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dolph R. Dawson, DMD,MS, Principal Investigator — University of Kentucky College of Dentistry; Jeff L. Ebersole, Ph.D, Study Chair — University of Kentucky College of Dentistry; M J Novak, Ph.D, Study Director — University of Kentucky College of Dentistry; Gilbert A. Boissonneault, Ph.D, Study Director — University of Kentucky Division of Clinical Nutrition
Locations (1):
- University of Kentucky College of Dentistry, Lexington, Kentucky, United States